CLINICAL TRIAL: NCT05580198
Title: Prognostic Markers of Post-Stroke Depression: A Single-center Prospective Observational Study
Brief Title: Prognostic Markers of Post-Stroke Depression (PROMoSD)
Acronym: PROMoSD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christos Krogias, Prof. Dr., Ruhr University of Bochum
Other Study IDs: 20-6862
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Acute Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- BRH+: Acute ischemic stroke patients with brainstem raphe hypoechogenicity.
  Interventions: Diagnostic Test: Transcranial sonography.
- BRH-: Acute ischemic stroke patients without brainstem raphe hypoechogenicity.
  Interventions: Diagnostic Test: Transcranial sonography.

INTERVENTIONS:
Diagnostic Test: Transcranial sonography. — Transcranial sonography examination to determine the brainstem raphe echogenicity.

SUMMARY:
Single-center prospective observational study investigating the association of brainstem raphe hypoechogenicity detected by transcranial sonography and post-stroke depression three months after an acute ischemic stroke.

DETAILED DESCRIPTION:
Post-stroke depression (PSD) is an important complication after a stroke. Despite significant limitations between studies of PSD risk factors, stroke severity or post-stroke disability, prior depressive episodes, and female sex are arguably the most well-known risk factors for developing PSD, although the predictive value of these factors is limited.

A hypoechogenic brainstem raphe (BR) detected by transcranial sonography (TCS) is associated with depressive symptoms in distinct diseases but is also common with approximately 25% of the non-depressed population in Europe. The primary aim of this study is to investigate the association between BR hypoechogenicity and PSD occurrence in a prospective observational study design.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke with the onset of symptoms within the past 14 days
* Diagnosis of AIS is confirmed by brain imaging, either computer tomography or magnetic resonance imaging

Exclusion Criteria:

* Insufficient transtemporal bone window for transcranial sonography examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who present with an acute ischemic stroke to the emergency department with the onset of symptoms within the past 14 days.
Sampling Method: Probability Sample
Enrollment: 105 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-11 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Post-stroke depression | 3 months
  PSD diagnosis was defined according to the fifth version of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V criteria) or by any new medication for anti-depressive indication during follow-up

SECONDARY OUTCOMES:
Severity of depressive symptoms | 3 months
  Measured by the Hamilton Depression Rating Scale (HRSD, minimum score: 0, maximum score: 52), with higher scores indicating greater severity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Christos Krogias, Prof., Principal Investigator — St. Josef-Hospital Bochum, Ruhr-University Bochum
Locations (1):
- St. Josef-Hospital Bochum, Bochum, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Richter D, Ebert A, Mazul-Wach L, Ruland Q, Charles-James J, Gold R, Tsivgoulis G, Juckel G, Krogias C. Prognostic markers of post-stroke depression (PROMoSD): study protocol of a prospective single-center observational study on raphe hypoechogenicity as a predictor of post-stroke depression. Neurol Res Pract. 2022 Dec 9;4(1):59. doi: 10.1186/s42466-022-00225-5. PMID 36494874